CLINICAL TRIAL: NCT04152551
Title: Effects of Bisphosphonates on OI-Related Hearing Loss: A Pilot Study
Brief Title: Effects of Bisphosphonates on OI-Related Hearing Loss
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: The New York Community Trust (Other); East River Medical Imaging (Unknown); Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: #2018-0700
Record Dates: First submitted 2019-10-18; First posted 2019-11-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-01

CONDITIONS: Osteogenesis Imperfecta
Keywords: hearing loss; bisphosphonate; skeletal dysplasia; brittle bone disorder; osteogenesis imperfecta; OI
MeSH Terms: conditions — Osteogenesis Imperfecta; Hearing Loss; Mucopolysaccharidosis IV; Brittle Bone Disorder | interventions — Risedronic Acid

STUDY DESIGN:
Intervention Model Description: 25 adults with type 1 OI and diagnosed hearing loss will be treated with oral risedronate.
  25 adults with type 1 OI will be enrolled into the control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Adult Treatment Arm (Experimental): Intervention treatment arm. Adults (18+ years) with type 1 OI. Must have at least mild hearing loss. Will receive Risedronate (35mg, 0-2x/week as clinically indicated) for duration of study. Changes in hearing, quality of life, and bone density will be monitored.
  Interventions: Drug: Risedronate Oral Tablet
- Child (Bisphosphonate Arm) (No Intervention): Observational (no investigational intervention) arm. Children (6-17 years) with any type of OI who are already receiving bisphosphonate treatment as standard of care treatment for orthopedic symptoms. Changes in hearing, quality of life, and bone density will be observed for the duration of the study.
- Child (Control Arm) (No Intervention): Observational arm. Children (6-17 years) with any type of OI who are not receiving bisphosphonate treatment. Changes in hearing, quality of life, and bone density will be observed for the duration of the study.
- Adult Control Arm (No Intervention): Observational arm. Adults (18+ years) with type 1 OI. Changes in hearing, quality of life, and bone density will be monitored.

INTERVENTIONS:
Drug: Risedronate Oral Tablet — Oral bisphosphonate
  Other Names: actonel
  Arms: Adult Treatment Arm

SUMMARY:
Osteogenesis Imperfecta-related hearing loss usually occurs in individuals with mild (type I) OI and is much earlier in onset than age-related hearing loss, with the majority of individuals experiencing some minor hearing loss in their 20s. Bisphosphonates have been successfully used to treat otosclerosis, a common cause of hearing loss similar to OI-related hearing loss. As many individuals with OI-related hearing loss also present with otosclerosis and because of their mechanistic similarities, the investigators propose studying the effects of bisphosphonate treatment on individuals diagnosed with both OI type I and hearing loss, thereby determining its effectiveness as a potential treatment for hearing loss.

The investigators will enroll 50 individuals diagnosed with type I OI and age 18-100. 25 adults will be enrolled into the treatment arm and receive bisphosphonate treatment (must have at least mild hearing loss), while 25 adults will be enrolled into the control arm. The investigators will enroll 25 children (6-17 years of age) diagnosed with OI who are currently receiving bisphosphonate treatment as part of their care for orthopedic symptoms. The investigators will also observe 25 children (6-17 years of age) diagnosed with OI who are NOT currently receiving bisphosphonate treatment. The study duration is 63 months (approximately 5 years). Enrollment is anticipated to begin in November 2019.

ELIGIBILITY:
Inclusion Criteria (Adult Treatment Arm):

* Diagnosis of OI type I
* Diagnosis of at least mild hearing loss (>20dB pure tone average) by audiogram testing
* 18+
* Vitamin D level > 30

Inclusion Criteria (Adult Control Arm):

* Diagnosis of OI type I

Inclusion Criteria (Child Observational Bisphosphonate Arm)

* Diagnosis of OI
* Age 6-17 years
* Currently receiving bisphosphonate treatment as standard of care

Inclusion Criteria (Child Observational No Treatment Arm)

* Diagnosis of OI
* Age 6-17 years
* NOT receiving bisphosphonate treatment and will not receive bisphosphonate treatment for the duration of the study

Exclusion Criteria (ALL ARMS):

* Family history of hearing-loss (not related to OI or occupational hearing loss)
* Pregnancy

Ages: 6 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Pure Tone Averages | Baseline, 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 months
  Average hearing thresholds at 250, 500, 1000, 2000, 3000, 4000, 8000 Hertz

SECONDARY OUTCOMES:
Speech Recognition Scores | Baseline, 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 months
  Lowest volume participant can hear and understand speech (decibels)
Word Recognition Scores | Baseline, 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 months
  Percent of words participants correctly repeat in word recognition test (%)
Hearing Handicap Inventory Raw Score | Yearly (Baseline, 12, 24, 36, 48, 60 months)
  Score 0-40. Lower score is better. Adults (self-reported)
Tinnitus Handicap Inventory Score | Yearly (Baseline, 12, 24, 36, 48, 60 months)
  Score 0-100. Lower score is better. Adults (self-reported).
Dizziness Handicap Inventory Score | Yearly (Baseline, 12, 24, 36, 48, 60 months)
  Score 0-100. Lower score is better. Adults (self-reported). Incidence and impact of vertigo in study population.
SF-36 Scale and Summary Scores | Yearly (Baseline, 12, 24, 36, 48, 60 months)
  Score 0-100. Higher score is better. Adults (self-reported) quality-of-life survey.
Pediatric Outcomes Data Collection Instrument (PODCI) Score | Yearly (Baseline, 12, 24, 36, 48, 60 months)
  Score 0-100. Lower score is better. Children (ages 6-10 years), parent-reported. Assessment of overall health and functioning.
Adolescent Outcomes Questionnaire Score | Yearly (Baseline, 12, 24, 36, 48, 60 months)
  Score 0-100. Lower score is better. Children (ages 11-17 years), parent- or self-reported. Assessment of overall health and functioning.
DEXA Z-score | Yearly (Baseline, 12, 24, 36, 48, 60 months)
  Higher score is better. Relative Bone Density
DEXA Bone Mineral Density | Yearly (Baseline, 12, 24, 36, 48, 60 months)
  Higher score is better. Bone Mineral Density (grams/centimeter^2)

CONTACTS AND LOCATIONS:
Overall Officials: Cathleen Raggio, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Dijk FS, Sillence DO. Osteogenesis imperfecta: clinical diagnosis, nomenclature and severity assessment. Am J Med Genet A. 2014 Jun;164A(6):1470-81. doi: 10.1002/ajmg.a.36545. Epub 2014 Apr 8. PMID 24715559
- [Background] Pillion JP, Vernick D, Shapiro J. Hearing loss in osteogenesis imperfecta: characteristics and treatment considerations. Genet Res Int. 2011;2011:983942. doi: 10.4061/2011/983942. Epub 2011 Dec 14. PMID 22567374
- [Background] Sillence D. Osteogenesis imperfecta: an expanding panorama of variants. Clin Orthop Relat Res. 1981 Sep;(159):11-25. PMID 7285446
- [Background] Swinnen FK, De Leenheer EM, Coucke PJ, Cremers CW, Dhooge IJ. Audiometric, surgical, and genetic findings in 15 ears of patients with osteogenesis imperfecta. Laryngoscope. 2009 Jun;119(6):1171-9. doi: 10.1002/lary.20155. PMID 19358256
- [Background] Berger G, Hawke M, Johnson A, Proops D. Histopathology of the temporal bone in osteogenesis imperfecta congenita: a report of 5 cases. Laryngoscope. 1985 Feb;95(2):193-9. doi: 10.1288/00005537-198502000-00014. PMID 3918222
- [Background] Vincent R, Wegner I, Stegeman I, Grolman W. Stapedotomy in osteogenesis imperfecta: a prospective study of 32 consecutive cases. Otol Neurotol. 2014 Dec;35(10):1785-9. doi: 10.1097/MAO.0000000000000372. PMID 24751750
- [Background] Plotkin LI, Weinstein RS, Parfitt AM, Roberson PK, Manolagas SC, Bellido T. Prevention of osteocyte and osteoblast apoptosis by bisphosphonates and calcitonin. J Clin Invest. 1999 Nov;104(10):1363-74. doi: 10.1172/JCI6800. PMID 10562298
- [Background] Rogers MJ, Frith JC, Luckman SP, Coxon FP, Benford HL, Monkkonen J, Auriola S, Chilton KM, Russell RG. Molecular mechanisms of action of bisphosphonates. Bone. 1999 May;24(5 Suppl):73S-79S. doi: 10.1016/s8756-3282(99)00070-8. No abstract available. PMID 10321934
- [Background] Drake MT, Clarke BL, Khosla S. Bisphosphonates: mechanism of action and role in clinical practice. Mayo Clin Proc. 2008 Sep;83(9):1032-45. doi: 10.4065/83.9.1032. PMID 18775204
- [Background] Kanzaki S, Ito M, Takada Y, Ogawa K, Matsuo K. Resorption of auditory ossicles and hearing loss in mice lacking osteoprotegerin. Bone. 2006 Aug;39(2):414-9. doi: 10.1016/j.bone.2006.01.155. Epub 2006 Mar 24. PMID 16564235
- [Background] Quesnel AM, Seton M, Merchant SN, Halpin C, McKenna MJ. Third-generation bisphosphonates for treatment of sensorineural hearing loss in otosclerosis. Otol Neurotol. 2012 Oct;33(8):1308-14. doi: 10.1097/MAO.0b013e318268d1b3. PMID 22935809
- [Background] Kang WS, Nguyen K, McKenna CE, Sewell WF, McKenna MJ, Jung DH. Measurement of Ototoxicity Following Intracochlear Bisphosphonate Delivery. Otol Neurotol. 2016 Jul;37(6):621-6. doi: 10.1097/MAO.0000000000001042. PMID 27153329
- [Background] Ting TH, Zacharin MR. Hearing in bisphosphonate-treated children with osteogenesis imperfecta: our experience in thirty six young patients. Clin Otolaryngol. 2012 Jun;37(3):229-33. doi: 10.1111/j.1749-4486.2012.02476.x. No abstract available. PMID 22708940
- [Background] Patel RM, Nagamani SC, Cuthbertson D, Campeau PM, Krischer JP, Shapiro JR, Steiner RD, Smith PA, Bober MB, Byers PH, Pepin M, Durigova M, Glorieux FH, Rauch F, Lee BH, Hart T, Sutton VR. A cross-sectional multicenter study of osteogenesis imperfecta in North America - results from the linked clinical research centers. Clin Genet. 2015 Feb;87(2):133-40. doi: 10.1111/cge.12409. Epub 2014 May 30. PMID 24754836